CLINICAL TRIAL: NCT04500548
Title: 3CI Study: Childhood Cancer Combination Immunotherapy. Phase Ib and Expansion Study of Nivolumab Combination Immunotherapy in Children, Adolescent and Young Adult (CAYA) Patients With Relapsed/Refractory Hypermutant Cancers
Brief Title: Testing the Combination of Two Immunotherapy Drugs (Nivolumab and Ipilimumab) in Children, Adolescent, and Young Adult Patients With Relapsed/Refractory Cancers That Have an Increased Number of Genetic Changes, The 3CI Study
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate accrual rate
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-05617; NCI-2020-05617 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PED-CITN-01 (Other: Cancer Immunotherapy Trials Network); PED-CITN-01 (Other: CTEP); P30CA015704 (NIH); UM1CA154967 (NIH)
Record Dates: First submitted 2020-08-04; First posted 2020-08-05 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Constitutional Mismatch Repair Deficiency Syndrome; Hematopoietic and Lymphoid Cell Neoplasm; Lynch Syndrome; Recurrent Lymphoma; Recurrent Malignant Solid Neoplasm; Recurrent Neuroblastoma; Recurrent Primary Central Nervous System Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Neuroblastoma; Refractory Primary Central Nervous System Neoplasm; Xeroderma Pigmentosum
MeSH Terms: conditions — Turcot syndrome; Hematologic Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis; Lymphoma; Neuroblastoma; Central Nervous System Neoplasms; Xeroderma Pigmentosum | interventions — Specimen Handling; Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose level -1 (nivolumab) (Experimental): PART I: Patients undergo collection of tissue samples for TMB level. Patients with elevated TMB may be eligible for Part II.
  PART II: Patients receive nivolumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biospecimen Collection; Biological: Nivolumab
- Dose level 1 (nivolumab, ipilimumab) (Experimental): PART I: Patients undergo collection of tissue samples for TMB level. Patients with elevated TMB may be eligible for Part II.
  PART II: Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive nivolumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for up to 23 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biospecimen Collection; Biological: Ipilimumab; Biological: Nivolumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of tissue samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
  Arms: Dose level 1 (nivolumab, ipilimumab)
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo

SUMMARY:
This phase Ib trial investigates the side effects of the combination of nivolumab and ipilimumab, and to see how well they work in treating patients with cancers that have come back (relapsed) or does not respond to treatment (refractory) and have an increased number of genetic changes. Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Tumor mutational burden (TMB) is the total amount of genetic changes or "mutations" found in tumor cells. Some studies in adults with cancer have shown that patients with a higher TMB (an increased number of genetic changes) are more likely to respond to immunotherapy drugs. There is also evidence that nivolumab and ipilimumab can shrink or stabilize cancer in adult patients with cancer. This study is being done to help doctors learn if the combination of nivolumab and ipilimumab can help children, adolescents, and young adults patients live longer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To confirm the safety and tolerability of nivolumab-based combination therapy in children, adolescent and young adult (CAYA) patients with relapsed/refractory hypermutant cancers (including solid tumors, central nervous system [CNS] tumors, neuroblastoma, and lymphoma).

Ia. To determine the tolerability, define and describe the toxicities, and determine the recommended phase 2 dose (RP2D) of nivolumab and ipilimumab combination therapy in CAYA patients with relapsed/refractory hypermutant cancers.

SECONDARY OBJECTIVE:

I. To assess objective overall response rate (ORR) to the nivolumab-based combination therapy in CAYA patients with relapsed/refractory hypermutant cancers within the confines of a Phase 1b study.

EXPLORATORY OBJECTIVES:

I. To assess clinical benefit rate (CBR) (objective response and stable disease for at least two [2] protocol reassessments), progression-free survival (PFS), and overall survival (OS) following nivolumab-based combination therapy in CAYA patients with relapsed/refractory hypermutant cancers.

II. To explore correlations between tumor genotype (including tumor mutation burden [TMB], specific gene mutations, etc.) and response to nivolumab-based combination therapy in CAYA patients with relapsed/refractory hypermutant cancers.

III. To discover biomarkers predicting response of hypermutant CAYA cancers undergoing PD-1 blockade including tumor neoantigen formation, specific T-cell receptor rearrangements (TCRR) of tumor infiltrating lymphocytes (TILs), and detailed characterization and activation of the immune infiltrations including the TILs.

IV. To explore the use of minimally invasive methods to monitor and predict response to immune checkpoint inhibition in hypermutant cancers including assessment of circulating tumor deoxyribonucleic acid (DNA) and circulating T-cells immunophenotypic profiling (differentiation markers, cytokines, etc.).

OUTLINE:

PART I: Patients undergo collection of tissue samples for TMB level. Patients with elevated TMB may be eligible for Part II.

PART II: Patients are assigned to 1 of 2 dose levels.

DOSE LEVEL 1: Patients receive nivolumab intravenously (IV) over 30-90 minutes and ipilimumab IV over 30 minutes on day 1. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive nivolumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for up to 23 cycles in the absence of disease progression or unacceptable toxicity.

DOSE LEVEL -1: Patients receive nivolumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 12 weeks for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* PART 1: Patients must have histologically or cytologically confirmed malignancy at the time of initial diagnosis, relapse, or recurrence. Patients must have recurrent or refractory cancer for which standard curative or palliative measures do not exist or are no longer effective

  * Patients with multiple concurrent and/or sequential neoplasms are eligible
  * Patients with central nervous system (CNS) tumors are eligible, except those with diffuse intrinsic pontine glioma
  * Patients with lymphoma are eligible; patients with leukemia are excluded
  * Chemotherapy-naive patients are eligible in cases where first-line therapy does not include chemotherapy (e.g., surgery only for ependymoma management)
* PART 1: Patients must have evidence of one or more of the following criteria in current or previous tumor:

  * Microsatellite instability (MSI-H)
  * Mutation causing functional loss of mismatch repair gene expression (MLH1, MSH2, MSH6, PMS2, EPCAM, MSH3)
  * Hypermutation in any tumor (including primary malignancy for patients with relapse or previous cancer diagnoses)
  * Functional mutation of POLE or POLD1 genes
  * A syndrome linked to hypermutant cancer predisposition such as congenital mismatch repair deficiency (CMMRD), Lynch syndrome, or xeroderma pigmentosum (XP) is also permitted
  * Other factors or sequencing evidence not listed above but which may be predictive of hypermutant cancer may be permitted after discussion with the protocol principal investigator
* PART 1: A tumor tissue specimen must be provided for molecular profiling, including TMB analysis. The specimen may be archival or prospective, from a medically necessary surgery, biopsy, or excision. Tissue will not be obtained solely for this trial. A specimen from the time of most recent relapse/progression is preferred, but not mandatory

  * Tissue is preferred. However, if necessary, previously extracted DNA may be used with the approval of the protocol principal investigator if extracted in a clinically certified laboratory and prepared in an Foundation Medicine Inc. (FMI), TMB assay-compatible manner
* PART 1: All patients and/or their parents or legally authorized representatives must have the ability to understand and the willingness to sign a written informed consent. Assent, where appropriate, will be obtained according to local policy. Patients with impaired decision-making capacity will not be excluded
* PART 2: Patients must have histologically or cytologically confirmed malignancy at the time of initial diagnosis, relapse, or recurrence. Patients must have recurrent or refractory cancer for which standard curative or palliative measures do not exist or are no longer effective

  * Patients with multiple concurrent and/or sequential neoplasms are eligible
  * Patients with CNS tumors are eligible, except those with diffuse intrinsic pontine glioma or bulky tumors
  * Patients with lymphoma are eligible (provided other criteria, such as bone marrow function, are met); patients with leukemia are excluded
  * Chemotherapy-naive patients are eligible in cases where first-line therapy does not include chemotherapy (e.g., surgery only for ependymoma management)
* PART 2: Patients must have measurable disease

  * Patients with neuroblastoma without measurable soft tissue but with iobenguane (MIBG) avid disease are eligible
  * Patients with bone marrow only disease are excluded
* PART 2: Patients must have confirmation of cancer with a TMB of >= 10 mutations (mut)/megabase (Mb) as determined by an next generation sequencing (NGS) targeted cancer gene panel performed by Foundation Medicine Inc. (FMI). Proof of TMB eligibility can be from Part 1 participation or a previously acquired FMI report
* PART 2: Patients must have recovered from the acute toxic effects of all prior anti-cancer therapies (with the exception of alopecia and lymphopenia)

  * Previous treatment with nivolumab and/or other anti-PD-1/PD-L1 inhibitors is permitted
  * Previous treatment with ipilimumab and/or other anti-CTLA-4 inhibitors is permitted
  * Previous treatment with combined anti-PD-1/PD-L1 and anti-CTLA-4 inhibitors is not be permitted
* PART 2: The following time periods apply for prior therapy. Patients must have:

  * Cytotoxic chemotherapy: At least 21 days prior to treatment initiation from the last dose of cytotoxic or myelosuppressive chemotherapy; at least 42 days if prior nitrosourea (such as lomustine, CCNU)
  * Hematopoietic growth factors: At least 7 days prior to treatment initiation from the last dose of short-acting growth factor; at least 14 days for long-acting
  * Anti-cancer agents not known to be myelosuppressive: At least 7 days prior to treatment initiation from the last dose
  * Interleukins, interferons, and cytokines (other than hematopoietic growth factors): At least 21 days prior to treatment initiation from the last dose
  * Antibodies: At least 21 days prior to treatment initiation from the last dose and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Radiotherapy: At least 14 days prior to treatment initiation from local radiotherapy; at least 150 days from total body irradiation (TBI), craniospinal radiotherapy, or radiation to >= 50% of the pelvis; at least 42 days from other substantial bone marrow radiation
  * Radiopharmaceutical therapy (e.g., 131I-MIBG): At least 42 days prior to treatment initiation from systemically administered radiopharmaceutical therapy
  * Autologous stem cell infusion including boost infusion: At least 42 days prior treatment initiation
  * Cellular therapy: At least 42 days prior to treatment initiation from any type of cellular therapy
* PART 2: Lansky play score >= 50 if =<16 years of age; Karnofsky performance scale >= 50 if =< 16 years of age. Patients unable to walk due to paralysis but who are using a wheelchair will be considered ambulatory for the purpose of assessing performance status
* PART 2: Peripheral absolute neutrophil count (ANC) >= 750/mm^3 (0.75 x 10^9/L)
* PART 2: Platelet count >= 75,000/mm^3 (75 x 10^9/L), transfusion independent, defined as not receiving platelet transfusions at least 7 days prior to treatment initiation
* PART 2: Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2; OR serum creatinine based on age/gender as follows:

  * Age: 1 to < 2 years; Maximum serum creatinine: 0.6 mg/dL; 53 umol/L (male); 0.6 mg/dL; 53 umol/L (female)
  * Age: 2 to < 6 years; Maximum serum creatinine: 0.8 mg/dL; 71 umol/L (male); 0.8 mg/dL; 71 umol/L (female)
  * Age: 6 to < 10 years; Maximum serum creatinine: 1 mg/dL; 88 umol/L (male); 1 mg/dL; 88 umol/L (female)
  * Age: 10 to < 13 years; Maximum serum creatinine: 1.2 mg/dL; 106 umol/L (male); 1.2 mg/dL; 106 umol/L (female)
  * Age: 13 to < 16 years; Maximum serum creatinine: 1.5 mg/dL; 133 umol/L (male); 1.4 mg/dL; 124 umol/L (female)
  * Age: >= 16 years; Maximum serum creatinine: 1.7 mg/dL; 150 umol/L (male); 1.4 mg/dL; 124 umol/L (female)
* PART 2: Bilirubin (sum of conjugated and unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* PART 2: Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 135 U/L (i.e., 3 x ULN). For the purposes of this study, the ULN for ALT (SGPT) is 45 U/L
* PART 2: No evidence of dyspnea at rest, no exercise intolerance due to pulmonary insufficiency, and pulse oximetry >= 92% while breathing room air
* PART 2: No signs or symptoms of heart failure in a patient who has no history of congestive heart failure, no prior exposure to cardiotoxic drugs, and no radiotherapy to the heart; OR shortening fraction of >= 27% or ejection fraction of >= 50% by echocardiogram
* PART 2: Serum lipase =< ULN at screening
* PART 2: Patients with treated CNS metastasis are eligible if there is no evidence of progression for at least 4 weeks after CNS-directed treatment as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT] scan) during screening

  * Patients with new or progressive CNS metastasis (active metastasis) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS-directed treatment is not required and is unlikely to be required for at least 6 weeks after treatment initiation, and a risk-benefit analysis (discussion) by the patient and investigator favors participation in the trial
* PART 2: Human immunodeficiency virus (HIV): Infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months prior to treatment initiation are eligible

  * Note: Routine screening for HIV status prior to enrollment is not required
* PART 2: Hepatitis B virus (HBV): Patients with evidence of chronic infection with undetectable viral load are eligible. Suppressive therapy, if indicated, is allowed

  * Note: Routine screening for HBV status prior to enrollment is not required
* PART 2: Hepatitis C virus (HCV): Infected patients currently on treatment with undetectable viral load are eligible. Patients with history of infection must have been treated and cured

  * Note: Routine screening for HCV status prior to enrollment is not required
* PART 2: Patients must provide a pre-treatment tumor tissue specimen (baseline sample) for correlative exploratory biology studies. The specimen may be archival or prospective, from a medically necessary surgery, biopsy, or excision. Tissue will not be obtained solely for this trial. A specimen from the time of most recent relapse/progression is preferred, but not mandatory. Submission of a representative sample from all available lesions (archival and prospective) is strongly encouraged. If available, residual tissue from Part 1 may be used to fulfill the baseline tissue sample requirement; however additional tissue may be required if residual tissue is insufficient
* PART 2: All patients and/or their parents or legally authorized representatives must have the ability to understand and the willingness to sign a written informed consent. Assent, where appropriate, will be obtained according to local policy. Patients with impaired decision-making capacity will not be excluded

Exclusion Criteria:

* PART 1: Patients with history of autoimmune disease
* PART 1: Patients with history of interstitial lung disease or pneumonitis are not eligible
* PART 1: Patients who have received solid organ transplant or allogenic stem cell transplant are not eligible
* PART 1: Patients who have been previously treated with a combination of anti-PD-1/PD-L1 and anti-CTLA-4 inhibitors are not eligible
* PART 2: Patients requiring systemic corticosteroids or other forms of immunosuppressive therapy within 7 days prior to treatment initiation are not eligible

  * Following treatment initiation, systemic corticosteroids or other forms of immunosuppressive therapy are permitted if administered for the treatment of toxicity, tumor flare, or pseudo-progression and can be tapered. In most cases study treatment must be held until the dose is tapered to 10 mg/day prednisone or equivalent. The protocol principal investigator must be consulted prior to resuming treatment
  * Physiologic corticosteroids up to 5 mg/day prednisone or equivalent are permitted
  * Topical, ocular, intra-articular, intra-nasal, inhaled corticosteroids are permitted
  * Patients with CNS tumors receiving steroids for intracranial mass effect must be able to discontinue these at least 7 days prior to treatment initiation
* PART 2: Patients who are receiving other anticancer agent(s) are not eligible
* PART 2: Patients who are receiving or have received any other investigational agent(s) within 14 days prior to treatment initiation are not eligible
* PART 2: Patients with CNS tumors with any of the following characteristics on imaging are not eligible:

  * Tumor with any evidence of uncal herniation or mass effect leading to severe midline shift
  * Tumor > 6 cm in single maximal dimension
  * Tumor that in the opinion of the investigator shows significant mass effect
* PART 2: Patients with uncontrolled intercurrent illness/condition that would limit compliance with the study requirements are not eligible. This includes, but is not limited to, ongoing active infection, symptomatic congestive heart failure (New York Heart Association class III or IV), unstable angina pectoris, cardiac arrhythmia, psychiatric illness/social situations
* PART 2: The study agents have the potential for teratogenic or abortifacient effects. Females of reproductive potential must have a negative serum pregnancy test within 72 hours prior to treatment initiation. Additional pregnancy tests (serum or urine) should be obtained during study participation in accordance with local standards and guidelines

  * Females of reproductive potential may not participate unless they have agreed to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of treatment, and as follows:

    * A period of 5 months after the last dose of nivolumab
    * A period of 3 months after the last dose of ipilimumab
  * Should a female patient become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform the investigator immediately
  * Due to the unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with the study agents, breastfeeding must be discontinued if the mother is treated on study
  * Males will not be required to use contraceptive measures
  * Note: Females of reproductive potential are defined as those who are past the onset of menarche and are not surgically sterile (i.e., bilateral salpingectomy, bilateral oophorectomy, complete hysterectomy)
* PART 2: Patients with history of autoimmune disease (such as autoimmune thyroid disease or inflammatory bowel disease) that has required systemic treatment within 2 years prior to treatment initiation are not eligible

  * Asymptomatic laboratory abnormalities (e.g., antinuclear antibody [ANA], rheumatoid factor, altered thyroid studies) are permitted in the absence of an autoimmune disorder diagnosis
  * Atopy-related conditions (e.g., asthma, allergic rhinitis, atopic dermatitis) are permitted
  * Replacement therapy (e.g., thyroxine, insulin, physiological corticosteroid replacement therapy) is not considered a form of systemic treatment
* PART 2: Patients with history of interstitial lung disease or pneumonitis are not eligible
* PART 2: Patients who have received solid organ transplant or allogenic stem cell transplant are not eligible
* PART 2: Patients with previous grade 4 life-threatening reaction or other adverse reaction that in the opinion of the investigator would preclude

Ages: 12 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days after last dose of study drug
  Graded by the revised National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0.

SECONDARY OUTCOMES:
Objective overall response rate (ORR) | Up to 1 year
  The portion of patients achieving complete response (iCR/CR) or partial response (iPR/PR). Response duration is measured from the time of initial response until documented disease progression.
Clinical benefit rate (CBR) | Up to 1 year
  The sum of the objective response (OR) and stable disease (iSD/SD) for at least two protocol reassessments periods.
Progression-free survival | From study entry until documented disease progression or death, assessed up to 1 year
Overall survival | From study entry or initial diagnosis until death from any cause, assessed up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Morgenstern, Principal Investigator — Cancer Immunotherapy Trials Network
Locations (9):
- United States (7):
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (2):
  • Informed Consent Form: PPED-CITN-01_A03ConsentPart1(Untracked).pdf (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT04500548/ICF_000.pdf
  • Informed Consent Form: PPED-CITN-01_A03ConsentPart2(Untracked).pdf (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT04500548/ICF_001.pdf